CLINICAL TRIAL: NCT04511936
Title: Microcurrent Stimulation Therapy for Dry Age-related Macular Degeneration (i-SIGHT): a Multicenter, Randomized, Double-masked, Clinical Device Trial
Brief Title: Microcurrent Stimulation for Dry Age-related Macular Degeneration
Acronym: i-SIGHT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-related delays.
Sponsor: i-Lumen Scientific, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILS-AMD-101
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Dry Age-related Macular Degeneration
Keywords: AMD; Dry AMD

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- i-Lumen AMD Active (Active Comparator)
  Interventions: Device: i-Lumen AMD
- i-Lumen AMD Sham (Sham Comparator)
  Interventions: Device: i-Lumen AMD Sham

INTERVENTIONS:
Device: i-Lumen AMD — Microcurrent stimulator
  Arms: i-Lumen AMD Active
Device: i-Lumen AMD Sham — Sham microcurrent stimulator
  Arms: i-Lumen AMD Sham

SUMMARY:
Evaluate the safety and efficacy of microcurrent stimulation therapy for patients with dry age-related macular degeneration.

DETAILED DESCRIPTION:
Multi-center, double-masked, randomized trial of microcurrent stimulation for the treatment of patients affected with dry age-related macular degeneration.

ELIGIBILITY:
Key Inclusion Criteria - Study Eye:

* Dry AMD diagnosis.

Key Exclusion Criteria - Study Eye:

* Wet AMD

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in best-corrected distance visual acuity (CDVA) at one month timepoint. | 1 Month

SECONDARY OUTCOMES:
Best-corrected distance visual acuity (CDVA) response rate at 1 month visit. | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Jackson, MD, Principal Investigator — King's College London

IPD SHARING:
Plan to Share IPD: No